CLINICAL TRIAL: NCT02341378
Title: A Multicenter, Single-blind, Phase 2A Clinical Trial to Evaluate the Efficacy and Safety of TissueGene-C, a Cell-mediated Gene Therapy, in Degenerative Arthritis Patients
Brief Title: Efficacy and Safety Study of TissueGene-C to Degenerative Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kolon Life Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TCG-K1-02
Record Dates: First submitted 2015-01-08; First posted 2015-01-19 (Estimated); Last update posted 2015-01-22 (Estimated); Status verified 2015-01

CONDITIONS: Degenerative Arthritis
Keywords: chondrocyte cells; Osteoarthritis; gene therapy
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TissueGene-C (Low dose) (Experimental): Single intra-articular injection to the damaged knee joint at a dose of 6.0 x 10^6 cells
  Interventions: Biological: TissueGene-C(Low dose)
- TissueGene-C (High dose) (Experimental): Single intra-articular injection to the damaged knee joint at a dose of 1.8 x 10^7 cells
  Interventions: Biological: TissueGene-C(High dose)

INTERVENTIONS:
Biological: TissueGene-C(Low dose) — TissueGene-C at 6.0x10^6 cells
  Arms: TissueGene-C (Low dose)
Biological: TissueGene-C(High dose) — TissueGene-C at 1.8x10^7 cells
  Arms: TissueGene-C (High dose)

SUMMARY:
To assess the efficacy and safety of the intra-articular injection of TissueGene-C in patients with degenerative arthritis of the knee

DETAILED DESCRIPTION:
TissueGene-C is a biological new drug which consists of non-transduced chondrocytes and transduced chondrocytes that express Transforming Growth Factor(TGF)-b1 to regenerate the damaged cartilage.

During the clinical trial Phase 2A, we compare low dose or high dose TissueGene-C in 6 months trial with 28 outpatients who have degenerative arthritis. The patients are randomized to two dose levels of TisssueGene-C by 1:1 ratio, and they are monitored and recorded for alleviating symptoms, sports activities, function of the knee, and the presence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 45 years or more
2. With grade 4 degenerative arthritis of the knee [based on the International Cartilage Repair Society(ICRS) evaluation criteria from the MRI results]
3. With less than 6 cm2major lesions
4. With major lesions (grade 4) concentrated in only one section of the knee and considered the main cause of the clinical symptoms
5. Unresponsive to conventional symptomatic treatment
6. Healthy and with no major physical examination, hematology, serum chemistry, and urine test findings and no significant medical history
7. Agreed to use an effective contraceptive method during the study period
8. Voluntarily agreed to participate in this study and signed the Informed Consent Form

Exclusion Criteria:

1. Abnormal screening laboratory test (hematology, serum, and urine test) findings
2. Took anti-inflammatory medications (prescribed or over-the-counter), including natural medicines, within 14 days before the injection of the investigational product
3. Took antirheumatic drugs (e.g., methotrexate or antimetabolites) within three months before enrollment in this study
4. Has a history of drug abuse within one year from the enrolment, or has positive results in the urine drug test or serum alcohol test at the screening visit
5. Received an injection in the target knee within two months before enrollment in this study
6. Pregnant or breastfeeding female
7. With another joint disease apart from degenerative arthritis (e.g., systemic rheumatic inflammatory disease associated with the knee or chondrocalcinosis, hemachromatosis, inflammatory arthritis, necrosis of the trochanter, Paget's disease adjacent to a joint in the femur or tibia, ochronosis, hemophilic arthropathy, infectious arthritis, Charcot's disease in the knee joint, villonodular synovitis, and synovial chondromas)
8. With a current infectious disease, including HIV or hepatitis
9. Has any of the following clinically significant diseases:

   * heart disease [e.g., myocardial infarction, arrhythmia, other serious heart disease, coronary artery bypass graft (CABG)]
   * kidney disease (e.g., chronic renal failure, glomerulonephritis)
   * liver disease (e.g., liver cirrhosis, fatty liver, acute or chronic liver disease)
   * endocrine disease (e.g., hyperthyroidism, hypothyroidism, thyroiditis, diabetes insipidus, Cushing's disease)
   * insulin-dependent diabetes mellitus
   * medical history of or current malignant tumor
   * In particular, the tumors that TissueGene-C may aggravate can be screened using the following tests:

     * Leukemia: White Blood Cell level in the hematology
     * Osteochondroma, Chondromas, Chondroblastoma, Chondromyxoid fibroma, Chondrosarcoma : Alkaline phosphatase level in the hematology
10. Participated in another clinical trial (using the investigational drug or a medical device) within 30 days before enrollment in this study
11. Considered by the investigator inappropriate for participation in this study

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-08; Primary Completion 2010-06 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Changes in IKDC Subjective Knee Evaluation | Week 0, 12 and 24
  Symptoms, sports activities, and function of the knee will be measured by the International Knee Documentation Committee (IKDC)

SECONDARY OUTCOMES:
Changes in WOMAC scores | Week 0, 12 and 24
  Pain, stiffness, and physical function of the knee will be measured by the Western Ontario and McMaster Universities(WOMAC)
Changes in 100 mm-VAS | Week 0, 12 and 24
  Pain of the knee will be measured by the 100mm Visual Analogue Scale (VAS)
Comparative Evaluation of Knee MRI | Week 0, 12 and 24
  Change in the Magnetic Resonance Images (MRI) scan results after the administration of TissueGene-C
Number of Participants with Adverse Events | Week 0, 2, 4, 12 and 24
  Allergic reaction, Injection site reaction , Infection in the injection site, Fibrosis, Fibrosis-deep connective tissue, Muscular/skeletal hypoplasia, TGF-β1 Enzyme-linked Immunosorbent Assay (ELISA) result, Polymerase Chain Reaction(PCR) for the vector DNA test results
Evaluation of Physical examination and laboratory tests | Week 0, 2, 4, 12 and 24
  Vital signs, Physical examination findings, Monitoring of the hematology, serum chemistry, and urine test results

CONTACTS AND LOCATIONS:
Overall Officials: Chul-won Ha, MD, PhD, Principal Investigator — Samsung Medical Center; Myung-chul Lee, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (3):
- South Korea (3):
  - Samsung Medical Center, Gangnam-gu, Seoul
  - Seoul National Univ. Hospital, Seoul
  - Asan Medical Center, Seoul

REFERENCES:
- [Derived] Ha CW, Cho JJ, Elmallah RK, Cherian JJ, Kim TW, Lee MC, Mont MA. A Multicenter, Single-Blind, Phase IIa Clinical Trial to Evaluate the Efficacy and Safety of a Cell-Mediated Gene Therapy in Degenerative Knee Arthritis Patients. Hum Gene Ther Clin Dev. 2015 Jun;26(2):125-30. doi: 10.1089/humc.2014.145. Epub 2015 Apr 17. PMID 25760423